CLINICAL TRIAL: NCT05454956
Title: Randomized, Double-Masked, Pilot Study Comparing the Safety and Efficacy of Two Dosing Regimens of TP-03 for the Treatment of Meibomian Gland Dysfunction in Patients With Demodex Lid Infestation
Brief Title: Pilot Study Comparing the Safety and Efficacy of Two Dosing Regimens of TP-03 for the Treatment of MGD
Acronym: Ersa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tarsus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRS-008
Record Dates: First submitted 2022-06-27; First posted 2022-07-12 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Meibomian Gland Dysfunction; Blepharitis; Demodex Infestation
Keywords: Demodex
MeSH Terms: conditions — Meibomian Gland Dysfunction; Blepharitis

STUDY DESIGN:
Intervention Model Description: Arm 1: Two doses of TP-03, 0.25% and one dose of TP-03 vehicle to maintain masking daily
  Arm 2: Three doses of TP-03, 0.25% daily
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment assignment (BID or TID) will be unknown to the study participant, investigators and site staff performing study assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BID Dosing (Experimental): TP-03, lotilaner ophthalmic solution, 0.25% administered topically twice a day and TP-03 vehicle administered once a day to maintain masking for approximately 85 days
  Interventions: Drug: TP-03; Drug: TP-03 Vehicle
- TID Dosing (Experimental): TP-03, lotilaner ophthalmic solution, 0.25% administered topically three times a day for approximately 85 days
  Interventions: Drug: TP-03

INTERVENTIONS:
Drug: TP-03 — TP-03, lotilaner ophthalmic solution, 0.25%, administered twice a day in participants in the BID dosing arm and three times a day in participants in the TID dosing arm
Drug: TP-03 Vehicle — Vehicle of TP-03 ophthalmic solution, administered once a day in participants in the BID dosing arm to maintain masking between arms
  Arms: BID Dosing

SUMMARY:
The purpose of this study is to compare the safety and efficacy of TP-03, 0.25%, an eyedrop, BID vs TID dosing regimens for the treatment of meibomian gland dysfunction in patients with Demodex lid infestation.

DETAILED DESCRIPTION:
This Phase 2a study is a randomized, two-arm, double-masked, multicenter, parallel pilot study to compare the safety and efficacy of two dosing regimens of TP-03, BID vs TID, for the treatment of meibomian gland dysfunction in patients with Demodex lid infestation. The primary objective of the study is to assess the safety and efficacy of two dosing regimens of TP-03, 0.25% from Day 1 to Day 85 in adult participants with meibomian gland dysfunction in the presence of Demodex infestation. Efficacy will be determined by assessing lower lid meibomian gland secretion, lid margin erythema, bulbar redness, tear breakup time, ocular surface staining, and dry eye symptoms. Safety will be determined by assessing adverse effects related to the treatment as well as evaluating any changes in visual acuity and slit lamp biomicroscopy from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to sign the informed consent and deemed capable of complying with the requirements of the study protocol
* Meets all of the following criteria in at least one eye: have more than 10 lashes with collarettes present on the upper lid; have the presence of one or more mites in the upper and lower lids; have evidence of meibomian gland dysfunction; have at least mild erythema of the lower lid; have a tear breakup time of less than 10 seconds; and have intact partial to full meibomian glands in at least 33% of the total meibomian gland area of the lower lid

Exclusion Criteria:

* Have used lid hygiene products within 7 days of Day 1 or unwilling to forego the use of lid hygiene products during the study
* Have used systemic antihistamines within 30 days of Day 1
* Have used artificial eyelashes, eyelash extensions or had other cosmetic eyelash or eyelid procedures within 7 days of Day 1 or be unwilling to forego their use during the study
* Contact lens wear within 7 days of Day 1 or unwilling to forego contact lens wear for the duration of the study
* Be pregnant or lactating at Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Shultz, MD, Principal Investigator — Mitchell C. Shultz, MD
Locations (5):
- United States (5):
  - Mitchell C. Shultz, MD, Northridge, California
  - Silverstein Eye Center, Kansas City, Missouri
  - Oculus Research, Cary, North Carolina
  - CORE Inc., Shelby, North Carolina
  - Medical Optometry America, New Freedom, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol stated up to 40 subjects to be enrolled. A total of 39 subjects were enrolled in the study which adhered to the protocol.
Groups:
- BID Dosing: TP-03, lotilaner ophthalmic solution, 0.25% administered topically twice a day and TP-03 vehicle administered once a day
- TID Dosing: TP-03, lotilaner ophthalmic solution, 0.25% administered topically three times a day
Period: Overall Study
Arm/Group | BID Dosing | TID Dosing
Started | 21 | 18
Completed | 20 | 18
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BID Dosing | TID Dosing | Total
Number analyzed (Participants) | 21 | 18 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (15.74) | 66.6 (13.13) | 63.7 (14.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 19 | 16 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 18 | 15 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 18 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs related (definitely or potentially) to treatment summarized by MedDRA preferred term.
Time Frame: 85 days
Measure: Count of Participants; unit: Participants
Arm/Group | BID Dosing | TID Dosing
Number analyzed (Participants) | 21 | 18
Participants | 1 | 1

2. Other Pre Specified Outcome: Change From Baseline in Lower Lid Meibomian Gland Secretion Score at Day 85
Description: For each of the 15 glands expressed, meibomian gland secretion characteristics were graded via slit lamp examination on a scale of 0 to 3 (0=worst, 3=best). Total meibomian gland secretion score is the sum of the grades for all 15 glands with a range from 0 to 45
Time Frame: Day 85 visit
Population: The analysis eye is defined as the eye that meets all eligibility criteria and was randomized per protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: analysis eye
Arm/Group | BID Dosing | TID Dosing
Number analyzed (Participants) | 20 | 18
Number analyzed (analysis eye) | 20 | 18
score on a scale | 10.5 (6.94) | 11.7 (7.89)

3. Other Pre Specified Outcome: Change From Baseline in Lid Margin Erythema (Upper Eyelid) at Day 85
Description: Erythema of the eyelid margin was assessed via slit lamp examination and graded on a scale of 0 (normal) to 3 (severe).
Time Frame: Day 85 visit
Population: The analysis eye is defined as the eye that meets all eligibility criteria and was randomized per protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: analysis eye
Arm/Group | BID Dosing | TID Dosing
Number analyzed (Participants) | 20 | 18
Number analyzed (analysis eye) | 20 | 18
score on a scale | -1.1 (0.85) | -1.0 (0.59)

ADVERSE EVENTS:
Time Frame: 200 days
Arm/Group | BID Dosing | TID Dosing
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/18
Other Adverse Events (participants affected / at risk) | 8/21 | 1/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BID Dosing (N=21) | TID Dosing (N=18)
Presyncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BID Dosing (N=21) | TID Dosing (N=18)
Conjunctivitis (Infections and infestations) | 1 | 1
Ocular discomfort (Eye disorders) | 1 | 0
Conjunctivochalasis (Eye disorders) | 1 | 0
Vitreous floaters (Eye disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0
Chemical burns of eye (Injury, poisoning and procedural complications) | 1 | 0
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
It is specified in the protocol that the data generated in this clinical trial, all related information and any materials containing such data and information are the exclusive property of Tarsus Pharmaceuticals, Inc. and are confidential to Tarsus Pharmaceuticals. Also, the investigator or other study-related personnel may not disclose to anyone or use any data, information or materials related to this clinical trial without the express written consent of Tarsus Pharmaceuticals.

DOCUMENTS (2):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT05454956/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT05454956/SAP_003.pdf